CLINICAL TRIAL: NCT00951574
Title: Prevention of Venous and Arterial Thromboembolism, in Cancer Patients Undergoing Chemotherapy, With a Low Molecular Weight Heparin (Nadroparin Calcium). A Randomized, Placebo-controlled, Double-blind, Multicenter Phase III Study.
Brief Title: Prevention of Venous and Arterial Thromboembolism, in Cancer Patients Undergoing Chemotherapy, With a Low Molecular Weight Heparin (Nadroparin Calcium)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DS/02/SELE/01
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: thromboembolism; cancer; chemotherapy; low-molecular-weight-heparin; nadroparin
MeSH Terms: conditions — Neoplasm Metastasis; Thromboembolism; Neoplasms | interventions — Nadroparin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline solution (Placebo Comparator): Pre-filled syringes of 0.4 ml, 1 subcutaneous injection/day (every 24 hours).
  Interventions: Drug: saline solution (placebo)
- nadroparin calcium (Experimental): Nadroparin calcium; Pre-filled syringes of 0.4 ml (3.800 anti-Xa IU), 1 subcutaneous injection/day (every 24 hours).
  Interventions: Drug: Nadroparin calcium

INTERVENTIONS:
Drug: Nadroparin calcium — Nadroparin calcium; Pre-filled syringes of 0.4 ml (3.800 anti-Xa IU), 1 subcutaneous injection/day (every 24 hours).
  Arms: nadroparin calcium
Drug: saline solution (placebo) — Pre-filled syringes of 0.4 ml , 1 subcutaneous injection/day (every 24 hours).
  Arms: saline solution

SUMMARY:
In this phase III, multicenter study, 1200 patients with lung, breast, gastrointestinal (stomach, colon-rectum, pancreas), ovarian or head and neck cancer undergoing chemotherapy will be randomly assigned (at the beginning of cytotoxic therapy) in a 2:1 ratio and in double-blind conditions to a treatment with subcutaneous low molecular weight heparin (nadroparin calcium, one injection/day) or placebo for the overall duration of chemotherapy or up to a maximum of 4 months (+/- 10 days).

ELIGIBILITY:
INCLUSION CRITERIA:

* both sexes;aged>18 years;
* suffering from different types of malignancies(lung, breast,gastric,colon- rectum,pancreatic,ovarian,head and neck cancer)undergoing systemic chemotherapy,
* having signed Informed Consent prior to initiation of any study procedure.

EXCLUSION CRITERIA:

* adjuvant and neo-adjuvant chemotherapy;
* objectively confirmed venous or arterial thromboembolism in the last three months;
* antithrombotic treatment for other indications;
* life expectancy of less than 3 months;
* Performance Status>2(ECOG);
* active bleeding or bleedings in the last four weeks requiring hospitalization,transfusion or surgical intervention;
* bleeding diathesis(prothrombin time<70% or activated partial thromboplastin time ratio>1.3),or platelet count<50x10^9/L;
* cerebrovascular hemorrhage in the last six months;
* known active gastric or duodenal ulcer;
* known cerebral metastasis;
* cerebral aneurysm;
* III-IV grade diabetic retinopathy;
* severe and uncontrolled hypertension(systolic blood pressure>180 mmHg or diastolic blood pressure>110 mmHg);
* chronic atrial fibrillation;
* acute endocarditis;
* acute pancreatitis;
* known hypersensitivity to unfractionated heparin or LMWH;
* previous occurrence of heparin-induced thrombocytopenia;
* renal impairment (dependent on dialysis or creatinine higher than 2.5mg%);
* liver insufficiency (alanine aminotransferase,aspartate aminotransferase,alkaline phosphatase levels>3 times the upper limit of the normal ranges and/or total bilirubin >3.0 mg/ml);
* pregnancy or childbearing potential without adequate contraception;
* treatment with other investigational drugs or patient inclusion in other clinical trials;
* patients who are unable to fulfill the study requirements in terms of visits/compliance to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1166 (Actual)
Dates: Start 2003-10; Primary Completion 2007-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of symptomatic venous and arterial thromboembolism, in patients with metastatic or locally advanced solid tumors undergoing chemotherapy | Events occurring during the four months of treatment plus 10 days

SECONDARY OUTCOMES:
Survival, at the end of study treatment | Events occurring during the four months of treatment plus 10 days
Response to chemotherapy | Events occurring during the four months of treatment plus 10 days
For patients with central venous catheters (CVC), complications of possible thrombotic origin, such as malfunction or requirement of CVC removal | Events occurring during the four months of treatment plus 10 days
Superficial thrombophlebitis of lower limbs | Events occurring during the four months of treatment plus 10 days
Asymptomatic thromboembolic events diagnosed during tests performed for other purposes | Events occurring during the four months of treatment plus 10 days
Safety (major bleeding, minor bleeding, other adverse events) | Events occurring during the four months of treatment plus 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Agnelli, MD, Study Chair — Internal and Vascular Medicine University of Perigia (Italy)
Locations (46):
- Italy (46):
  - Medical Oncology Department, Fabriano, Ancona
  - Medical Oncology Department Oncology Institute, Bari, Bari
  - Medical Oncology Unit, Bergamo, Bergamo
  - Medical Oncology Department, Treviglio, Bergamo
  - Medical Oncology Department - Bellaria Hospital, Bologna, Bologna
  - Medical Oncology Department - Businco Hospital, Cagliari, Cagliari
  - Medical Oncology Department University of Cagliari, Cagliari, Cagliari
  - Medical Oncology Department, Catanzaro, Catanzaro
  - Medical Oncology Department, Cosenza, Cosenza
  - Medical Oncology Department, Cremona, Cremona
  - Medical Oncology Department, Ferrara, Ferrara
  - Medical Oncology Department Careggi Hospital, Florence, Firenze
  - Casa Sollievo dell Sofferenza, San Giovanni Rotondo, Foggia
  - Cancer institute of Romagna, Forlì, Forlì
  - Medical Oncology Department, Latina, Latina
  - Medical Oncology Department, Lecce, Lecce
  - Medical Oncology Department, Lucca, Lucca
  - Medical Oncology Department, Taormina, Messina
  - Medical Oncology Department, Legnano, Milano
  - University Bicocca, Milan, Milano
  - Medical Oncology Department Fatebenefratelli Hospital, Milan, Milano
  - Medical Oncology Department Policlinico, Milan, Milano
  - Gynecology Oncology INT, Milan, Milano
  - Medical Oncology Department San Carlo Hospital, Milan, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Medical Oncology Department, Camposampiero, Padova
  - Medical Oncology Department Istituto Oncologico Veneto, Padua, Padova
  - Medical Oncology Department, Palermo, Palermo
  - Salvatore Maugeri Foundation, Pavia, Pavia
  - Medical Oncology Department, Città di Castello, Perugia
  - Medical Oncology Department, Perugia, Perugia
  - Medical Oncology Department, Todi, Perugia
  - Hematology and Oncology Department, Piacenza, Piacenza
  - Medical Oncology Department - University of Pisa, Pisa, Pisa
  - Medical Oncology Department, Ravenna, Ravenna
  - Medical Oncology Department, Reggio Emilia, Reggio Emilia
  - Medical Oncology Department - S Filippo Hospital, Roma, Roma
  - Medical Oncology Department Regina Elena Institute, Roma, Roma
  - Medical Oncology Department 3 Regina Elena Cancer Institute, Rome, Rome
  - Onco-gynecology Department - Catholic University, Rome, Rome
  - Medical Oncology Department, Sassari, Sassari
  - Medical Oncology Department, Terni, Terni
  - Medical Oncology Department San Luigi Hospital, Orbassano, Torino
  - Oncology Department Molinette Hospital, Torino, Torino
  - Medical Oncology Department, Varese, Varese
  - Medical Oncology Department, Viterbo, Viterbo

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Barni S, Labianca R, Agnelli G, Bonizzoni E, Verso M, Mandala M, Brighenti M, Petrelli F, Bianchini C, Perrone T, Gasparini G. Chemotherapy-associated thromboembolic risk in cancer outpatients and effect of nadroparin thromboprophylaxis: results of a retrospective analysis of the PROTECHT study. J Transl Med. 2011 Oct 20;9:179. doi: 10.1186/1479-5876-9-179. PMID 22013950
- [Derived] Agnelli G, Gussoni G, Bianchini C, Verso M, Mandala M, Cavanna L, Barni S, Labianca R, Buzzi F, Scambia G, Passalacqua R, Ricci S, Gasparini G, Lorusso V, Bonizzoni E, Tonato M; PROTECHT Investigators. Nadroparin for the prevention of thromboembolic events in ambulatory patients with metastatic or locally advanced solid cancer receiving chemotherapy: a randomised, placebo-controlled, double-blind study. Lancet Oncol. 2009 Oct;10(10):943-9. doi: 10.1016/S1470-2045(09)70232-3. Epub 2009 Aug 31. PMID 19726226